CLINICAL TRIAL: NCT03815370
Title: A Non-Traumatic Binder for Temporary Abdominal Wall Closure (ABRO) Multicentre Trial
Brief Title: A Non-Traumatic Binder for Temporary Abdominal Wall Closure
Acronym: ABRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-249
Record Dates: First submitted 2017-11-22; First posted 2019-01-24 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Abdominal Trauma; Abdominal Injury; Abdominal Infection; Abdominal Sepsis; Abdominal Abscess; Abdominal Aneurysm; Abdominal Compartment Syndrome; Peritonitis
Keywords: Abdominal trauma/injury; Abdominal sepsis/infection; Open Abdomen; Abdominal binder; Abthera; VAC; ABRO
MeSH Terms: conditions — Abdominal Injuries; Intraabdominal Infections; Abdominal Abscess; Aortic Aneurysm, Abdominal; Intra-Abdominal Hypertension; Peritonitis; Wounds and Injuries; Infections

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to compare usual care (vacuum or non-vacuum methods for temporary coverage of the OA) versus usual care plus the new abdominal binder device called ABRO™.
Masking Description: It is impossible for the participant or anyone within the patients circle of care to be blinded in this study, as it is clear if the abdominal binder is on the participant or not. There is no way to blind in this interventional study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Placebo Comparator): The current approach for temporary coverage of abdomen is called "vacuum assisted techniques (VAT)". This technique requires the use of vacuum-assisted drainage to remove blood or watery fluid from a wound or operative site.
  Interventions: Device: Placebo Comparator: Usual Care
- Device: ABRO™Binder Arm (Experimental): Intervention is the usual care (listed above) plus a novel new abdominal binder device called ABRO™
  Interventions: Device: Experimental: ABRO™ Binder Arm

INTERVENTIONS:
Device: Experimental: ABRO™ Binder Arm — ABRO™ is an abdominal device designed to be positioned superficially on the abdominal skin of patients managed with the Open Abdomen strategy. The device is comprised of two rigid plates to stabilize the abdominal muscles thus preventing buckling of these. Another element of this novel device is the circumferential dynamic retainer (CDR). This one is passed behind the patient's back to provide more stability to the muscles in the abdomen keeping them in position to prevent lateral movement of them.
  Arms: Device: ABRO™Binder Arm
Device: Placebo Comparator: Usual Care — The current approach for temporary coverage of abdomen is called "vacuum assisted techniques (VAT)". This technique requires the use of vacuum-assisted drainage to remove blood or watery fluid from a wound or operative site.
  Arms: Usual Care

SUMMARY:
At the end of most abdominal operations, the fascial layer is closed by stitching edges of the wound together. However, because of logistic and/or technical reasons or the patient's critical condition, the surgeon is forced to leave the abdomen open.

The current approach for temporary coverage of abdomen is vacuum assisted techniques (VAT). This technique requires the use of vacuum-assisted drainage to remove blood or watery fluid from a wound or operative site. Although this is the most successful and commonly used procedure, there are some limitations to this method. For example, VAT have little effect on preventing lateral movement of the wound edges. Therefore, VAT it is not the ideal procedure in aiding surgeons to closed the abdomen.

The purpose of this study is to compare usual care (vacuum or non-vacuum methods for temporary coverage of the OA) versus usual care plus a novel new abdominal binder device called ABRO™ that may aid in the closure of patients who undergo open abdomen closure procedures.

DETAILED DESCRIPTION:
At the end of most abdominal operations the fascial layer is closed primarily. However, because of logistic, physiological and or anatomical reasons, the surgeon needs to leave the abdomen open. In those circumstances, attempts to close the abdomen could potentially lead to unnecessary damage to the abdominal wall fascia, intra-abdominal hypertension, abdominal compartment syndrome and abdominal wall dehiscence post-operatively.

The use of the "open abdomen" (OA) in the post-operative period is not uncommon. Currently, three important trends provide grounds for increased use of this surgical strategy:

* Lifesaving surgical procedures in severely injured trauma patients.
* Surgical procedures performed in patients with non-traumatic surgical emergencies
* Abdominal catastrophes in elderly patients with pre-existing medical conditions. The OA is not a new strategy in the surgeon's armamentarium. A recent publication retrieved more than 1300 articles over the last 25 years relative to the management of the OA, published in the English language.5 However, the precise incidence of the OA is unknown. Nonetheless, hospitals around the world, particularly those that receive trauma victims, have an OA rate of 1-5% among their most critically ill surgical patients.

This lifesaving surgical strategy does not come without a price. The mortality rate of an OA is approximately 30%. There is also a wide range of complications linked to this procedure. The OA exposes large surface area of the body to the environment increasing fluid losses. Maintenance of adequate fluid and nutritional status of the patient are challenging in this setting.

Furthermore, the exposed abdominal cavity also poses greater risk for local contamination from external sources that could ultimately result in sepsis. Impaired abdominal wall function interferes with ventilatory mechanics. Consequently, patients with OA are prone to respiratory complications. However, the most dreaded complication of an OA is the formation of an enteroatmospheric fistula (EF). The incidence of EF is approximately 11-15%, and increases with time. Patients who have an OA for more than 8 days have an incidence of ECF as high as 25%, caused mainly by damage to the exposed bowel. Management this complication is extremely challenging, very costly, and carries a mortality rate of 36-64%.

In consideration of the foregoing considerations, early closure of the OA is undoubtedly the most effective way to prevent complications linked to this lifesaving surgical strategy. One of the most important barriers to early closure of the OA is lateral retraction of the fascial wound edges. Retraction presents as early as three days post-operatively, involves all layers of the abdominal wall and ultimately results in loss of domain. Moreover, generalized edema, atrophy and contraction of the abdominal muscles also contribute to a progressively larger defect in the fascia.Another important problem is "buckling" of the rectus abdominal muscles resulting in a "diamond" shape defect in the fascial that is very difficult to close.

Management of the OA prior to definitive closure call for temporary closure techniques. The three main objectives of temporary closure techniques are to prevent injury to the bowel, manage fluid loss from the abdominal cavity, and ultimately to facilitate primary closure. Early closure is dependent on technical factors and patients' underlying clinical condition. Despite all efforts to facilitate primary fascial closure, this condition is successfully achieved only in approximately 60% of the cases.

Currently, vacuum assisted techniques (VAT) are the most frequent, and arguably the most efficacious method for temporary coverage of the OA. Furthermore, VAT are particularly useful in the management of edema fluid, gastrointestinal and peritoneal secretions. Despite these important benefits, VAT provide minimal support to prevent lateral retraction of the abdominal wall fascial edges. Indeed, vacuum closure devices are not able to brace the abdominal wall and prevent lateralization of the rectus muscles even with maximum negative pressure. Moreover, excessive negative pressure applied to the abdominal cavity could potentially provoke severe injury to the intra-abdominal organs and interfere with physiologic functions.

Devices applied surgically to the abdominal wall are more effective in preventing lateral retraction of the fascial edges. However, these devices are stitched through the skin, subcutaneous tissue, muscle, and fascial layers. These stitches frequently cut through the aforementioned tissues because of the high pressure at the suture sites produced by counteracting forces. The resulting wounds encompass all layers of the abdominal wall including the fascia. Another important drawback of devices that require a surgical procedure for application is the need for frequent trips to operating room for assessment and potential adjustments. Furthermore, technical limitations inherit to surgically applied temporary closure devices result in undesirable delay for the initial placement. A recent report showed that the mean time from the primary operation to placement of the temporary closure device was 9.5 days.16 This is dangerously close to the critical period of EF formation and loss of abdominal domain.

Interim analysis of the data obtained from the initial randomized clinical trial to investigate the original prototype of the non-traumatic binder for abdominal wall closure (ABROTM) described in this protocol showed promising results (n=20 patients). The utilization of the original prototype of the ABROTM device resulted in 80% primary fascial closure rate compared to only 50% when VAT alone was employed. All patients (n=10) subjected to the application of the original prototype of the ABROTM device had their abdomen closed by primary fascial suture, without component separation or mesh. The ABROTM prototype resulted in greater than 65% reduction in the maximum width and the area of the fascial defects at 4 ± 1 days post-operative, whereas VAT alone resulted in a 5% increase. Moreover, interim analysis of the data showed that there were no complications from the use of the prototype of the ABROTM device. Therefore, it is anticipated that the use of the new ABROTM device in the proposed multicentre randomized controlled trial may have several advantages compared to preexisting methods for closure of the OA

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients, managed with the OA strategy.
* 16 years of age or older

Exclusion Criteria:

* Patients who are pregnant
* Loss of any portion of the abdominal wall that could preclude primary closure
* Burn patients
* BMI greater than 40 kg/m2

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Total number of patients who experience complete abdominal closure with sutures without the use of mesh and/or component separation. | Outcome measures will record when closure of the abdomen takes place up to 11 days after randomization.
  The primary outcome will measure the total number of patients who experience complete abdominal closure with sutures without the use of mesh and/or component separation.

CONTACTS AND LOCATIONS:
Overall Officials: Joao Rezende-Neto, MD, Principal Investigator — Unity Health Toronto
Locations (4):
- Canada (4):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - St. Michael's Hospital, Toronto, Ontario